CLINICAL TRIAL: NCT00269724
Title: Open-Label Safety And Dose Conversion/Determination Study of OROS® Oxybutynin Chloride for Urge Urinary Incontinence
Brief Title: A Study to Evaluate the Safety and Efficacy of OROS® Oxybutynin Chloride for the Treatment of Urge Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR005971
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-04

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; oxybutynin; OROS®
MeSH Terms: conditions — Urinary Incontinence

INTERVENTIONS:
Drug: OROS® oxybutynin

SUMMARY:
The purpose of this study is to is to evaluate the safety and efficacy of OROS® oxybutynin chloride in patients being treated for urge urinary incontinence. Oxybutynin is an antispasmodic, anticholinergic medication for the treatment of the symptoms of overactive bladder.

DETAILED DESCRIPTION:
Urinary incontinence refers to the involuntary loss of urine in sufficient amounts to be considered a social or health problem. It is under-reported and under-treated as patients are often ashamed and embarrassed to discuss their condition and clinicians may also fail to ask patients about incontinence. This is a multi-center, open-label study including dose conversion and dose determination to evaluate the safety of OROS® oxybutynin chloride at a clinically acceptable dose. There are three study periods: Run-in, Dose Conversion/Determination, and Maintenance. During the 1-week Run-in Period, baseline incontinence, urinary frequency, and health related quality-of-life data are collected. During the Dose Conversion/Determination Period, any previous urge urinary incontinence medications are discontinued and each patient is started on OROS® oxybutynin chloride. The dose is titrated to a clinically acceptable dose in 5-mg increments at 7 ± 3 day intervals to a possible maximum dose of 30 mg/day. The clinically acceptable dose is defined as either the minimum effective dose (i.e., the dose at which the patient has no incontinent episodes for the last 2 days of the dosing interval) or the dose providing the best balance between symptomatic improvement and side effects. Patients taking immediate-release oxybutynin at enrollment started dose titration on OROS® oxybutynin chloride at a dose equal to their immediate-release oxybutynin dose; all others started at 5 mg per day OROS® (oxybutynin chloride). After the clinically acceptable dose is established, the patient continues for an additional week at that dose to confirm that it is appropriate. Then the patient enters the 12-week Maintenance Period that evaluates whether the urge urinary incontinence reduction that is achieved by the beginning of maintenance has persisted. The primary outcome of the study is an evaluation of the safety of OROS® oxybutynin chloride. Safety assessments include the incidence of adverse events, physical examination and medical history, clinical laboratory tests, urinalysis, electrocardiograms (ECGs), vital signs, and the Physician's Anticholinergic Effects Assessment (P-ACEA), an assessment completed by the physician if severe or intolerable anticholinergic effects occur.

OROS® oxybutynin chloride (5 mg and 10 mg systems): One to five systems taken orally per day (5 mg per day to a maximum of 30 mg per day) as a single morning dose. The duration of the Maintenance Period of the study is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-neurogenic urge urinary incontinence, neurogenic urge urinary incontinence, or mixed urge urinary incontinence with a clinically significant urge component
* Patients currently taking medications for urge urinary incontinence (that are listed in the protocol) including immediate-release oxybutynin chloride, or patients not currently taking medication for urge urinary incontinence who have had at least 6 urge urinary incontinence episodes during the 1-week Run-in Period
* Patients who are able to differentiate incontinent episodes associated with urgency from incontinent episodes not associated with urgency when recording incontinent episodes in the diary
* Patients who are in good general health prior to study participation, without significant bacteria or fewer than 10 WBC/hpf on urinalysis, or a negative urine culture
* Patients agreeing that a medically acceptable and effective birth control method will be used by the patient and partner throughout the study and for one week following the end of the study-drug treatment

Exclusion Criteria:

* Patients with known treatable genitourinary conditions that may cause incontinence (e.g., urinary tract infection, prostatitis, urinary tract obstruction, bladder tumor, bladder stone, prostate cancer)
* Patients with narrow-angle glaucoma or untreated narrow anterior chamber angles obstructive uropathy, partial or complete obstruction or narrowing of the gastrointestinal tract, paralytic ileus, intestinal atony, colitis or myasthenia gravis
* Patients with known allergy or hypersensitivity to oxybutynin chloride, or with clinically significant medical problems or other organ abnormality or pathology for whom, administration of oxybutynin chloride would present undue risk
* Male patients who have had prostate surgery less than six months before study enrollment or any history of prostate cancer
* Patients who have been treated with anticholinergic medications for urge urinary incontinence and have been found to be not responsive to these treatments, and patients who are at significant risk of developing complete urinary retention if placed on an anticholinergic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 1997-03; Study Completion 1997-09

PRIMARY OUTCOMES:
Incidence of adverse events; Results from Physician's Anticholinergic Effects Assessment (P-ACEA)

SECONDARY OUTCOMES:
Change from Week 1 to Week 12 of Maintenance Period in: Urge urinary incontinence episodes per week; Urinary incontinence episodes per week; Void frequency per week

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — Alza Corporation, DE, USA

REFERENCES:
- See also: Open-label safety and dose conversion/determination study of OROS® (oxybutynin chloride) for urge urinary incontinence — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=98&filename=CR005971_CSR.pdf